CLINICAL TRIAL: NCT04632108
Title: A 1/2 Phase Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of ASKB589 in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu Aosaikang Pharmaceutical Co., Ltd. (Industry)
Collaborators: Jiangsu Aosaikang Biopharmaceutical Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASK-LC-B589-I/II
Record Dates: First submitted 2020-11-05; First posted 2020-11-17 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Malignant Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ASKB589 Injection (Experimental): Experimental: ASKB589 Injection ASKB589 Injection treatment. This phase 1/II trial will include two stages, a dose escalation stage and an expansion stage.
  Interventions: Drug: ASKB589 Injection

INTERVENTIONS:
Drug: ASKB589 Injection — ASKB589 Injection with dose escalation stage of 0.3mg/kg up to 20mg/kg,as well as dose expansion stage with recommended dose level from dose escalation stage.

SUMMARY:
This is an open label Phase 1/2 study, the purpose of the trial is to assess the safety, tolerability, pharmacokinetics, and antitumor activity of ASKB589 in patients suffering from advanced or metastatic solid tumors. Patients with gastric cancer/gastroesophageal junction adenocarcinoma and pancreatic cancer are preferred.

ELIGIBILITY:
Inclusion Criteria:

1. According to RECIST 1.1 criteria, all patients must have at least one measurable lesion, and the tumor lesions must be accurately measured in at least one dimension, and lesions previously treated with radiotherapy or local therapy are only evaluated as non-target lesions. Bone metastatic lesions are not considered as measurable lesions;
2. ECOG performance status (PS) 0-1;
3. The results of the laboratory tests must meet all the following criteria:

（1）Haemoglobin≥9 g/dL；platelet count≥ 100 × 109/L；absolute neutrophil count≥ 1.5 × 109/L；

（2）Albumin≥ 3.0g/dL；total bilirubin ≤ 1.5 times the upper limit of normal (ULN)；aspartate transaminase and alanine aminotransferase≤ 2.5 times ULN if no demonstrable liver metastases ( ≤5 times ULN in the presence of liver metastases);

（3）Creatinine clearance≥ 50ml/min；

（4）Prothrombin time, international normalized ratio, and activated partial thromboplastin time≤1.5×ULN (except for patients receiving anticoagulant therapy)

4.Life expectancy of at least 3 months;

5.Patients who are supposed to be enrolled into the monotherapy dose escalation study must meet all the following criteria:

1. Patients of either gender, aged from 18 years old to 70;
2. Patients with histologically or cytologically confirmed diagnosis of advanced unresectable or metastatic malignant solid tumor, for whom have no standard therapy or have no access to standard therapy for various reasons.

6.Patients who are supposed to be enrolled into the monotherapy dose expansion study must meet all the following criteria:

1. Patients of either gender, aged ≥ 18 years old；
2. Patients with histologically or cytologically confirmed diagnosis of advanced unresectable or metastatic gastric cancer, gastroesophageal junction adenocarcinoma and pancreatic cancer, for whom have no standard therapy or have no access to standard therapy for various reasons, and that tumor tissue samples are CLDN18.2 positive detected by central laboratory (medium-high expression)；
3. Other tumor types with good potential benefits will be included according to the results of the clinical results of same target products (CLDN18.2-positive tumors).

7.Patients who are supposed to be enrolled into the dose escalation of ASKB589 combined with chemotherapy should meet all the following criteria:

1. Patients of either gender, aged from 18 years old to 70.
2. Patients with gastric cancer, gastroesophageal junction adenocarcinoma and pancreatic cancer who are tolerant to CAPOX, GEM+Nab-P chemotherapy.
3. Patients with gastric cancer, gastroesophageal junction adenocarcinoma who are intolerant to anti-human epidermal growth factor receptor 2 (anti-HER2) drug therapy.
4. Other tumor types with good potential benefits will be included according to the results of mono-therapy dose expansion and the clinical results of same target products.

8.Patients who are supposed to be enrolled into the dose expansion of ASKB589 combined with chemotherapy should meet all the following criteria:

1. Patients of either gender, aged ≥ 18 years old.
2. Patients with gastric cancer, gastroesophageal junction adenocarcinoma and pancreatic cancer who are tolerant to CAPOX, GEM+Nab-P chemotherapy, and that tumor tissue samples are CLDN18.2 positive detected by central laboratory.
3. Patients with gastric cancer, gastroesophageal junction adenocarcinoma that who are intolerant to anti-HER2 drug therapy.
4. Other tumor types with good potential benefits will be included according to the results of this study and the clinical results of same target products.

Exclusion Criteria:

1. Patients have a history of severe allergic reactions to monoclonal antibodies or are intolerance to monoclonal antibodies, or those who are allergic to experimental drug and any component of the drug.
2. Patients have received a treatment of whole blood or blood component transfusion or various growth factor treatments within 14 days prior to enrollment.
3. Patients have received anti-tumor therapy within 14 days prior to enrollment，including but not limited to radiotherapy, chemotherapy, targeted therapy, treatment with herbal medications or other treatments that have known antitumor activity . Patients who have undergone palliative radiotherapy for bone metastases and whose acute toxicity has returned to normal can be selected;
4. Patients have received systemic immunosuppressive therapy（such as systemic corticosteroids）within 14 days prior to enrollment. However, patients using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30mg per day of hydrocortisone or 10mg per day of prednisone) are allowed；patients are allowed to receive a single dose of systemic corticosteroids treatment；
5. Patients have participated in other clinical trials within 28 days prior to enrollment; patients who have participated monoclonal antibody clinical trials within 2 months prior to sign written informed consent form also cannot participate in this trial；
6. Patients have received major surgical operation within 28 days prior to enrollment or schedule to perform major surgery during the period of this clinical trial;
7. Patients have gastrointestinal diseases such as gastrinoma, duodenitis, gastric ulcer, duodenal ulcer, pancreatitis or upper gastrointestinal hemorrhage, caused by nonmalignant tumor (gastric cancer, gastroesophageal junction adenocarcinoma and pancreatic cancer)withinwithin 3 months prior to enrollment；Patients have gastric inlet and outlet obstruction or suspected obstruction within 1 months prior to enrollment；
8. Known to have irritable bowel syndrome, ulcerative colitis, Crohn's disease, gastric outlet obstruction, etc., or any other causes that can cause long-term chronic nausea,persistent repeated vomiting or diarrhea, and uncontrolled or severe gastrointestinal bleeding;
9. Have a history of diagnosed neurological or mental disorders, including epilepsy or dementia;
10. Patients with any other malignant tumors within the past 5 years, cured cervical carcinoma in situ, basal cell, or squamous cell skin cancer are not included;
11. Known active central nervous system (CNS) metastasis or suspected cancerous meningitis;
12. Uncontrollable third-space effusion in clinical practice, which is deemed unsuitable for enrollment by the researchers;
13. Patients currently suffering from diseases that affect intravenous injection and venous blood sampling;
14. Patients suffering from major cardiovascular diseases, including:

（1）Congestive heart failure (defined as New York Heart Association Class III or IV), myocardial infarction, unstable angina, coronary angioplasty, stenting, coronary artery bypass graft, cerebrovascular accident (CVA) or hypertensive crisis within 6 months before the first drug treatment；

（2）History of clinically significant ventricular arrhythmia (such as sustained ventricular tachycardia, ventricular fibrillation or torsade de pointes)；

（3）Patients have an abnormality in the 12-lead electrocardiogram (ECG) including a Fridericia's corrected QT interval (QTcF) greater than 450 milliseconds (ms) (males) or greater than 470 ms (females).

（4）History or family history of congenital long QT syndrome；

（5）Cardiac arrhythmias requiring anti-arrhythmic drug therapy (patients suffering from atrial fibrillation >1 month before the first administration of drug can be selected according to the condition of patients);

（6）Left ventricular ejection fraction <50%；

15.Pregnant or lactating women; or women of childbearing age who have a positive blood pregnancy test during screening period; or women of childbearing age and their spouses who are unwilling to take effective contraceptive measures during the period of this clinical trial and within 6 months after the end of the clinical trial;

16.Patients who are not meet the inclusion criteria based on the judgment of investigator；

17.Patients included in dose-escalation and expansion study of combined chemotherapy should also exclude:

1. Patients with gastric cancer, gastroesophageal junction adenocarcinoma who are allergic, intolerant or contraindicated to any other components of capecitabine and oxaliplatin.
2. Patients with pancreatic cancer who are allergic, intolerant or contraindicated any components of gemcitabine and albumin bound paclitaxel for injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with serious adverse events (SAE) as assessed by CTCAE v5.0 | up to 21 days following last dose
  An SAE is defined as any untoward medical occurrence that, at any dose: a.) Results in death; b.) Is life-threatening; c.) Requires inpatient hospitalization or prolongation of existing hospitalization; d.) Results in persistent or significant disability/incapacity; e.) Is a congenital anomaly/birth defect; f.) Other important medical events; The number of participants who experience an SAE will be presented.
The incidence and case number of DLT (Dose Limiting Toxicity) during observation period | up to 21 or 28 days following first dose
  DLT is short for Dose Limiting Toxicity，dose-limiting describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment.
Number of participants with adverse events as assessed by CTCAE v5.0 | up to 21 days following last dose
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be presented.
Maximum Tolerated Dose (MTD） | up to 21 or 28 days following first dose
  The MTD was defined as the highest dose of ASKB589 not causing DLT in more than 33% of patients in the first treatment cycle.
The recommended dose | from date of treatment start until data cut-off, up to 2 years
  The recommended dose will be determined during the dose escalation and dose expansion stage of the study.
Objective response rate | from date of treatment start until disease progression,date of death or withdrawal from study,whichever came first, up to 2 years
  Evaluation of objective response rate assessed by response evaluation criteria in solid tumors version 1.1(RECIST 1.1)

SECONDARY OUTCOMES:
Pharmacokinetics:maximum Plasma Concentration [Cmax] | Up to 21 days after injection
  Serum samples will be collected for Cmax analysis.
Pharmacokinetics:time to maximum observed plasma concentration (Tmax) | Up to 21 days after injection
  Serum samples will be collected for Tmax analysis.
Pharmacokinetics:elimination rate constant（Kel） | Up to 21 days after injection
  Serum samples will be collected for Kel analysis.
Pharmacokinetics:terminal elimination half life (T1/2) | Up to 21 days after injection
  Serum samples will be collected for T1/2 analysis.
Pharmacokinetics:apparent volume of distribution (Vz/F) | Up to 21 days after injection
  Serum samples will be collected for Vz/F analysis.
Pharmacokinetics:Area Under Curve (AUC) | Up to 21 days after injection
  Serum samples will be collected for AUC analysis.
Pharmacokinetics: Mean ResidenceTime（MRT） | Up to 21 days after injection
  Serum samples will be collected for MRT analysis.
Pharmacokinetics: plasma clearance rate (CL) | Up to 21 days after injection
  Serum samples will be collected for CL analysis.
Pharmacokinetics: steady-state peak concentration (Css_max) | Up to 21 days after injection
  Serum samples will be collected for Css_max analysis.
Pharmacokinetics: time to steady-state peak concentration (Tss_max) | Up to 21 days after injection
  Serum samples will be collected for Tss_max analysis.
Pharmacokinetics: minimum value of steady plasma drug concentration（Css_min） | Up to 21 days after injection
  Serum samples will be collected for Css max analysis.
Evaluation of immunogenicity | from date of treatment start until data cut-off, up to 2 years
  Incidence of anti-drug antibodies (ADA)
Objective response rate（ORR） | from date of treatment start until disease progression,date of death or withdrawal from study,whichever came first, up to 2 years
  Evaluation of objective response rate assessed by RECIST 1.1
disease control rate（DCR） | from date of treatment start until disease progression,date of death or withdrawal from study,whichever came first, up to 2 years
  Evaluation of Disease control rate assessed by RECIST 1.1
Duration of Response（DOR） | from date of treatment start until disease progression,date of death or withdrawal from study,whichever came first, up to 2 years
  Duration of response assessed by RECIST 1.1
Progression free survival（PFS） | from date of treatment start until the date of disease progression or until death due to any causes, up to 2 years.
  Progression of tumor will be measured by RECIST v1.1
Overall survival（OS） | from the date of treatment start until the documented date of death from any cause，up to 2 years.
  defined as the time from the date of treatment start until date of death due to any cause

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing cancer hospital, Beijing, Beijing Municipality
  - Linyi cancer hospital, Linyi, Shandong

IPD SHARING:
Plan to Share IPD: No